CLINICAL TRIAL: NCT01150435
Title: Driving Ability of Drug Dependant Patients in Maintenance Therapy
Status: Completed | Type: Observational
Sponsor: Hummel, Christiane (Individual)
Collaborators: Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Christiane Hummel, Christiane Hummel
Other Study IDs: Hummel 2010-1
Record Dates: First submitted 2010-06-23; First posted 2010-06-25 (Estimated); Last update posted 2010-06-25 (Estimated); Status verified 2010-06

CONDITIONS: Driving Ability

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Drug screen Urin
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Maintenance Medication D, S- Methadon
- Maintenance Medication S- Methadon
- Buprenorphine
- Buprenorphine+ Naloxone

SUMMARY:
"Mobility" is a contributing factor in today's society. Drug dependence displays not only a medical but also an economic problem: Especially for an intended reintegration of a drug dependant patient in maintenance therapy the possession of a driving licence could be decisive for a job allocation and therefore the intended reintegration to society.

Subject of this study was to verify if patients under substitution therapy with R, S- Methadone, S- Methadone, Buprenorphine and Buprenorphine plus Naloxone are just as fit to drive a car as a non drug dependent person.

For this investigation we compared 121 drug dependent patients in stable maintenance therapy for a minimum of two years without consumption of any other psychotropic substances than their maintenance drug (including THC) with non- drug dependant subjects of the same gender, age and level of education.

This is the largest study on this topic worldwide. The neuro- cognitive working order was tested by means of the "Vienna Test System" an objective, reliable and valid test quantifying reaction time, attention efficiency, concentration, maximum resilience and orientation. Current use of any other psychotropic substance or alcohol just as any serious illness (including psychiatric diseases, except for an effectively treated depression) lead to exclusion from this study.

ELIGIBILITY:
Inclusion Criteria:

* Drug dependent patients in stable maintenance therapy for a minimum of two years without consumption of any other psychotropic substances than their maintenance drug (including THC)
* Written agreement on attending this study after full clarification
* majority

Exclusion Criteria:

* Patients, who do not approve or are not able to approve, to this study
* Patients, who are not legally competent
* Patients in emergency situations
* Patients under age
* Consumption of any other psychotropic substances than the maintenance drug
* Severe illnesses p.e. malignant diseases, serious psychiatric illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: drug dependent patients in stable maintenance therapy
Sampling Method: Non-Probability Sample
Enrollment: 121 (Actual)
Dates: Start 2008-02; Primary Completion 2010-04 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Gilg, Proffessor, Study Director — Institut für Rechtsmedizin München
Locations (1):
- Institut für Rechtsmedizin, Munich, Baveria, Germany